CLINICAL TRIAL: NCT01322685
Title: Development and Application of Rapid Nucleic Acid Diagnostic Kits for Clinical Specimens
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Kuo-Sheng Hung, Department of Neurosurgery, WanFang Hospital
Other Study IDs: 99042
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Tuberculosis; Lung Cancer
Keywords: Tuberculosis; Lung cancer
MeSH Terms: conditions — Tuberculosis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Health Group
- Tuberculosis Group: Tuberculosis or lung cancer group

SUMMARY:
The purpose of this study is to study the Development and Application of Rapid Nucleic Acid Diagnostic Kits for Clinical Specimens. Subjects are divided into two groups which are health group and Tuberculosis or lung cancer group in order to compare with the difference.

ELIGIBILITY:
Inclusion Criteria:

* Health group: between 17 to 90 years old
* Tuberculosis group: people who are tuberculosis or lung cancer patients and between 17 to 90 years old

Exclusion Criteria:

* Women subjects are before or after the period within two days

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health people Tuberculosis or lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Sheng Hung, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan